CLINICAL TRIAL: NCT02918565
Title: Mechanisms for Alcohol Treatment Change [MATCH] Study
Acronym: MATCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Maria Pacella, Research Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STUDY19050262; R01AA023650 (NIH)
Record Dates: First submitted 2016-09-23; First posted 2016-09-29 (Estimated); Results first posted 2023-12-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Alcohol Consumption
MeSH Terms: conditions — Alcohol Drinking | interventions — Ethanol

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Drinking Cognition Feedback (DCF) (Experimental): 12 weeks of interactive text messaging focused on providing feedback related only to pre-weekend drinking cognitions (plans, desire to get drunk).
  Interventions: Behavioral: Drinking Cognition Feedback (DCF)
- Alcohol Risk Feedback (ARF) (Experimental): 12 weeks of interactive text messaging focused on providing feedback related only to post-weekend alcohol consumption (max drinks consumed on any occasion over the weekend).
  Interventions: Behavioral: Alcohol Risk Feedback (ARF)
- Adaptive Goal Support (AGS) (Experimental): 10 weeks of interactive text messaging focused on providing adaptive goal support (based on running average of max drinks consumed).
  Interventions: Behavioral: Adaptive Goal Support (AGS)
- COMBO (Experimental): 12 weeks of interactive text messaging incorporating features of DCF, ARF and AGS.
  Interventions: Behavioral: COMBO
- Control (No Intervention): 12 weeks of text message assessments without any feedback

INTERVENTIONS:
Behavioral: Drinking Cognition Feedback (DCF) — 12 weeks of interactive text messaging focused on providing feedback related only to pre-weekend drinking cognitions (plans, desire to get drunk).
  Arms: Drinking Cognition Feedback (DCF)
Behavioral: Alcohol Risk Feedback (ARF) — 12 weeks of interactive text messaging focused on providing feedback related only to post-weekend alcohol consumption (max drinks consumed on any occasion over the weekend).
  Arms: Alcohol Risk Feedback (ARF)
Behavioral: Adaptive Goal Support (AGS) — 12 weeks of interactive text messaging focused on providing adaptive goal support (based on running average of max drinks consumed).
  Arms: Adaptive Goal Support (AGS)
Behavioral: COMBO — 12 weeks of interactive text messaging incorporating features of DCF, ARF and AGS.
  Arms: COMBO

SUMMARY:
A 5-arm randomized trial to determine what components of a text message intervention are necessary to reduce hazardous drinking among young adults and mechanisms through which these changes occur.

DETAILED DESCRIPTION:
Young adults ages 18-25 have high rates of hazardous alcohol use and alcohol-related consequences. The Emergency Department (ED) provides an important opportunity to identify young adult hazardous drinkers who could benefit from interventions. A Text Message (TM) intervention was shown to reduce alcohol consumption among young adult ED patients, showing durable effects over 9-months. The TM intervention uses behavior change techniques with the largest effect sizes in an alcohol intervention meta-analysis: "goal commitment" and "self-monitoring", along with real-time "feedback". However, the unique effect of these ingredients, and mechanisms (processes occurring within the individual) through which they operate to reduce drinking remain unclear, a critical gap addressed by this project. Young adult ED patients (ages 18-25) who screen positive for hazardous drinking will be recruited to participate in a randomized trial to determine how best to help individuals reduce hazardous drinking. All participants will be asked to complete web-based surveys at baseline, 12 and 24 weeks after enrollment, complete brief psychomotor tasks weekly for 14 weeks, and respond to text messages each Thursday and Sunday for the next 12 weeks. Those randomized to the TM interventions will additionally receive feedback on their text reports. The four TM intervention arms are: (1) Drinking Cognition Feedback (DCF), (2) Alcohol Risk Feedback (ARF), (3) Adaptive Goal Support (AGS) and (4) a combination of DCF, ARF, and AGS=COMBO). Study results have implications for designing efficient mobile interventions, and developing a dynamic theory of behavior change.

ELIGIBILITY:
Inclusion Criteria:

* total score of >2 for women or >3 for men on the AUDIT-C
* at least 1 binged drinking episode in the prior 30 days

Exclusion Criteria:

* no cell phone with text messaging
* have been diagnosed with an alcohol or substance use disorder
* pregnant or planning pregnancy
* taking medicine for a psychiatric disorder (including depression, anxiety)
* taking any medicine that could interact with alcohol

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1131 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2021-11-22 (Actual); Study Completion 2021-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Suffoletto, MD MS, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center Emergency Department, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified dataset provided upon request

REFERENCES:
- [Derived] Chung T, Suffoletto B, Bhurosy T. Which intervention works for whom: Identifying pre-treatment characteristics that predict who will benefit from a specific alcohol text message intervention from a randomized trial. J Subst Use Addict Treat. 2025 Jan;168:209562. doi: 10.1016/j.josat.2024.209562. Epub 2024 Nov 4. PMID 39505110
- [Derived] Bae SW, Suffoletto B, Zhang T, Chung T, Ozolcer M, Islam MR, Dey AK. Leveraging Mobile Phone Sensors, Machine Learning, and Explainable Artificial Intelligence to Predict Imminent Same-Day Binge-drinking Events to Support Just-in-time Adaptive Interventions: Algorithm Development and Validation Study. JMIR Form Res. 2023 May 4;7:e39862. doi: 10.2196/39862. PMID 36809294
- [Derived] Suffoletto B, Field M, Chung T. Attentional and approach biases to alcohol cues among young adult drinkers: An ecological momentary assessment study. Exp Clin Psychopharmacol. 2020 Dec;28(6):649-658. doi: 10.1037/pha0000343. Epub 2019 Dec 30. PMID 31886700

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | COMBO | Adaptive Goal Support (AGS) | Alcohol Risk Feedback (ARF) | Drinking Cognition Feedback (DCF) | Control
Started | 220 | 213 | 232 | 224 | 242
Completed | 213 | 202 | 221 | 216 | 231
Not Completed | 7 | 11 | 11 | 8 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | COMBO | Adaptive Goal Support (AGS) | Alcohol Risk Feedback (ARF) | Drinking Cognition Feedback (DCF) | Control | Total
Number analyzed (Participants) | 220 | 213 | 232 | 224 | 242 | 1131
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.8 (2.2) | 22.2 (2.0) | 22.1 (2.1) | 22.3 (2.1) | 22.1 (2.0) | 22.1 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 145 | 143 | 163 | 156 | 168 | 775
  Male | 75 | 70 | 69 | 68 | 74 | 356
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 19 | 17 | 14 | 28 | 97
  Not Hispanic or Latino | 201 | 194 | 215 | 210 | 214 | 1034
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 6 | 1 | 3 | 0 | 0 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 76 | 81 | 82 | 86 | 95 | 420
  White | 116 | 112 | 132 | 123 | 126 | 609
  More than one race | 13 | 14 | 11 | 9 | 14 | 61
  Unknown or Not Reported | 9 | 5 | 4 | 6 | 7 | 31
Any tobacco use [Number; unit: participants] | 123 | 117 | 120 | 117 | 105 | 582
Impulsivity score [Mean (Standard Deviation); unit: units on a scale] — Participants completed the Short Urgency, Premeditation, Perseverance, Sensation seeking, and Positive urgency (S-UPPS-P) scale. 20 items rated on a four-point Likert scale: (1) disagree strongly, (2) disagree some, (3) agree some, and (4) agree strongly. Five scales were computed by adding the 4 items corresponding to each scale: (1) negative urgency (NU), (2) positive urgency (PU), (3) sensation seeking (SS), (4) lack of perseveration (PE), and (5) lack of premeditation (PR). Range of total impulsivity (summary) score 20 to 80 with higher values representing more impulsivity.
  units on a scale | 41.4 (7.4) | 41.9 (6.7) | 41.3 (6.9) | 41.3 (6.9) | 41.4 (7.7) | 41.5 (7.1)

OUTCOME MEASURES:

1. Primary Outcome: Number of Binge Drinking Days
Description: Measured by the # days on the Timeline Followback Calendar that a male reported 5+ drinks or a female reported 4+ drinks
Time Frame: 12 weeks after starting intervention
Population: CCA
Measure: Mean (Standard Deviation); unit: days
Arm/Group | COMBO | Adaptive Goal Support (AGS) | Alcohol Risk Feedback (ARF) | Drinking Cognition Feedback (DCF) | Control
Number analyzed (Participants) | 169 | 175 | 192 | 180 | 201
days | 2.3 (3.3) | 2.6 (4.2) | 2.9 (4.3) | 3.0 (4.3) | 3.4 (4.2)

2. Secondary Outcome: Drinks Per Drinking Day
Description: drinks per drinking day = mean drinks divided by the number of days with any alcohol consumption using the 30-day TLFB Calendar.
Time Frame: 12 weeks after starting intervention
Measure: Mean (Standard Deviation); unit: drinks/day
Arm/Group | COMBO | Adaptive Goal Support (AGS) | Alcohol Risk Feedback (ARF) | Drinking Cognition Feedback (DCF) | Control
Number analyzed (Participants) | 169 | 175 | 192 | 180 | 201
drinks/day | 2.9 (2.5) | 2.9 (2.0) | 3.2 (2.1) | 3.0 (2.2) | 3.5 (2.2)

3. Secondary Outcome: Count of Participants With Any Binge Drinking Day
Description: Using the Timeline Followback Calendar, any male participant reported one or more days with 5+ drinks or a female with one or more days with 4+ drinks are coded=1; otherwise participant is coded=0
Time Frame: 12 weeks after starting intervention
Measure: Count of Participants; unit: Participants
Arm/Group | COMBO | Adaptive Goal Support (AGS) | Alcohol Risk Feedback (ARF) | Drinking Cognition Feedback (DCF) | Control
Number analyzed (Participants) | 169 | 175 | 192 | 180 | 201
Participants | 95 | 110 | 119 | 115 | 144

4. Secondary Outcome: Brief Young Adult Alcohol Consequences Questionnaire Score
Description: Brief Young Adult Alcohol Consequences Questionnaire (B-YAACQ). The B-YAACQ is a 24-item measure of alcohol- related problems that utilizes a dichotomous (present or absent) scoring format. Sum of items 1-48. Higher scores (count of items marked as 'present') on the B-YAACQ not only indicate a wider variety but also reflect a more severe pattern of alcohol-related problems.
Time Frame: 12 weeks after starting intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | COMBO | Adaptive Goal Support (AGS) | Alcohol Risk Feedback (ARF) | Drinking Cognition Feedback (DCF) | Control
Number analyzed (Participants) | 169 | 175 | 192 | 180 | 201
score on a scale | 4.1 (4.7) | 4.4 (5.1) | 5.0 (5.1) | 4.7 (5.3) | 5.6 (5.5)

ADVERSE EVENTS:
Time Frame: 6-months
Arm/Group | COMBO | Adaptive Goal Support (AGS) | Alcohol Risk Feedback (ARF) | Drinking Cognition Feedback (DCF) | Control
All-Cause Mortality (participants affected / at risk) | 0/220 | 0/213 | 0/232 | 0/224 | 0/242
Serious Adverse Events (participants affected / at risk) | 0/220 | 0/213 | 0/232 | 0/224 | 0/242
Other Adverse Events (participants affected / at risk) | 0/220 | 0/213 | 0/232 | 0/224 | 0/242

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-01): https://cdn.clinicaltrials.gov/large-docs/65/NCT02918565/Prot_SAP_000.pdf